CLINICAL TRIAL: NCT05987982
Title: Mouth Odor as a Precision Care Indicator for Preventing Pneumonia Among Middle-aged and Older Adults With Oral Frailty
Brief Title: Mouth Odor on Preventing Pneumonia by Oral Frailty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chen, Yen-Chin, Vice Head Nurse and Clinical Assistant Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-ER-111-452
Record Dates: First submitted 2023-07-18; First posted 2023-08-14 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Breathing, Mouth; Pneumonia; Frailty
Keywords: mouth odor; pneumonia; oral bacteria; oral frailty; oral management rehabilitation
MeSH Terms: conditions — Mouth Breathing; Pneumonia; Frailty | interventions — Exercise; Oral Hygiene; Dental Care Team

STUDY DESIGN:
Intervention Model Description: 1. Oral management group: oral exercises and oral care.
  2. Oral care group: oral hygiene.
  3. Routine group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group with oral management (Experimental): The investigators taught and monitored patients or caregivers to oral health care plus oral exercises such as salivary glands massage methods after meals and before sleep.
  Interventions: Procedure: Oral exercises and oral hygiene
- Group with oral care (Experimental): The investigators taught and monitored patients or caregivers to do oral care after meals and before sleep.
  Interventions: Procedure: Oral care
- Group with standard of care (No Intervention): Only provided oral care education.

INTERVENTIONS:
Procedure: Oral exercises and oral hygiene — The patients will be required to perform oral exercises and maintain oral hygiene twice a day. The investigators will assess their oral frailty, oral bacteria, oral odor, and other related clinical care data on the following time points: day 1 of hospitalization, day 3 of hospitalization, the day of discharge, one week after discharge, and one month after discharge.
  Arms: Group with oral management
Procedure: Oral care — The patients will be required to maintain oral hygiene twice a day. The investigators will assess their oral frailty, oral bacteria, oral odor, and other related clinical care data on the following time points: day 1 of hospitalization, day 3 of hospitalization, the day of discharge, one week after discharge, and one month after discharge.
  Arms: Group with oral care

SUMMARY:
This research plan aims to first collect data on the oral function and oral hygiene status of the elderly population in the community and to understand the normal model of oral frailty among the older adults in the community. Subsequently, a comparison will be made between the oral status of hospitalized patients and the community-dwelling elderly population. The goal is to verify whether oral odor can be used as an objective biological indicator following intervention.

DETAILED DESCRIPTION:
The first stage will aim to examine the relationships between the level of oral frailty and pneumonia-associated pathogens, as well as to establish a mouth odor database among community-dwelling people; The second stage will compare the differences of the level of oral frailty, pneumonia associated pathogens, and mouth odor between 144 middle-aged and older healthy people and 160 hospitalization patients. The third stage will confirm whether the mouth odor is an effective biological maker to show the changes of oral frailty, pneumonia-associated pathogens, and mouth odor after oral management rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old,
* Alert and oriented,
* With sufficient comprehension and cooperation,
* Willing to participate in oral assessment.

Exclusion Criteria:

* Patients who score below 5 on the General Practitioner Assessment of Cognition (GPCOG),
* Patients with oral treatments such as oral cancer treatment,
* Patients with oral treatments such as periodontal disease treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Clearance of pneumonia associated oral bacteria | The first day of admission (baseline)
  The investigators collected tongue specimens from participants for bacterial isolation and identification. The participants' specimens were collected using an eswab and sent for bacterial culture within 2 hours. Bacterial colonies were quantified (CFU/ml). To observe the variation caused by the number of bacteria, measurements were taken again after the intervention. The investigators assessed the clearance of bacteria based on the baseline.
Clearance of pneumonia associated oral bacteria | Day 3 of admission
  The investigators collected tongue specimens from participants for bacterial isolation and identification. The participants' specimens were collected using an eswab and sent for bacterial culture within 2 hours. Bacterial colonies were quantified (CFU/ml). To observe the variation caused by the number of bacteria, measurements were taken again after the intervention. The investigators assessed the clearance of bacteria based on the baseline.
Clearance of pneumonia associated oral bacteria | Discharge day
  The investigators collected tongue specimens from participants for bacterial isolation and identification. The participants' specimens were collected using an eswab and sent for bacterial culture within 2 hours. Bacterial colonies were quantified (CFU/ml). To observe the variation caused by the number of bacteria, measurements were taken again after the intervention. The investigators assessed the clearance of bacteria based on the baseline.
Clearance of pneumonia associated oral bacteria | 1-week after discharge day
  The investigators collected tongue specimens from participants for bacterial isolation and identification. The participants' specimens were collected using an eswab and sent for bacterial culture within 2 hours. Bacterial colonies were quantified (CFU/ml). To observe the variation caused by the number of bacteria, measurements were taken again after the intervention. The investigators assessed the clearance of bacteria based on the baseline.
Clearance of pneumonia associated oral bacteria | 1-month after discharge day
  The investigators collected tongue specimens from participants for bacterial isolation and identification. The participants' specimens were collected using an eswab and sent for bacterial culture within 2 hours. Bacterial colonies were quantified (CFU/ml). To observe the variation caused by the number of bacteria, measurements were taken again after the intervention. The investigators assessed the clearance of bacteria based on the baseline.
oral frailty measures (oral functions) | The first day of admission (baseline)
  The investigators measured seven items for patients to identify oral frailty including 1) the number of teeth, 2) masticatory ability, 3) difficulty making the "ta" sound, 4) tongue pressure, 5) abnormal swallowing pressure, and 6) tongue coating index (TCI), 7) oral dryness. Oral frailty was determined into three groups: non-oral frailty, 0 points; pre-oral frailty, 1-2 points; and oral frailty, ≥ 3 points.
oral frailty measures (oral functions) | Day 3 of admission
  The investigators measured seven items for patients to identify oral frailty including 1) the number of teeth, 2) masticatory ability, 3) difficulty making the "ta" sound, 4) tongue pressure, 5) abnormal swallowing pressure, and 6) tongue coating index (TCI), 7) oral dryness. Oral frailty was determined into three groups: non-oral frailty, 0 points; pre-oral frailty, 1-2 points; and oral frailty, ≥ 3 points.
oral frailty measures (oral functions) | Discharge day
  The investigators measured seven items for patients to identify oral frailty including 1) the number of teeth, 2) masticatory ability, 3) difficulty making the "ta" sound, 4) tongue pressure, 5) abnormal swallowing pressure, and 6) tongue coating index (TCI), 7) oral dryness. Oral frailty was determined into three groups: non-oral frailty, 0 points; pre-oral frailty, 1-2 points; and oral frailty, ≥ 3 points.
oral frailty measures (oral functions) | 1-week after discharge day
  The investigators measured seven items for patients to identify oral frailty including 1) the number of teeth, 2) masticatory ability, 3) difficulty making the "ta" sound, 4) tongue pressure, 5) abnormal swallowing pressure, and 6) tongue coating index (TCI), 7) oral dryness. Oral frailty was determined into three groups: non-oral frailty, 0 points; pre-oral frailty, 1-2 points; and oral frailty, ≥ 3 points.
oral frailty measures (oral functions) | 1-month after discharge day
  The investigators measured seven items for patients to identify oral frailty including 1) the number of teeth, 2) masticatory ability, 3) difficulty making the "ta" sound, 4) tongue pressure, 5) abnormal swallowing pressure, and 6) tongue coating index (TCI), 7) oral dryness. Oral frailty was determined into three groups: non-oral frailty, 0 points; pre-oral frailty, 1-2 points; and oral frailty, ≥ 3 points.
Oral odor | The first day of admission (baseline)
  A participant was requested to exhale two gas sampling gas for testing. The investigators uesd an E-nose to identify the participants' odor. To assess the variation of oral odor after different interventions.
Oral odor | Day 3 of admission
  A participant was requested to exhale two gas sampling gas for testing. The investigators uesd an E-nose to identify the participants' odor. To assess the variation of oral odor after different interventions.
Oral odor | Discharge day
  A participant was requested to exhale two gas sampling gas for testing. The investigators uesd an E-nose to identify the participants' odor. To assess the variation of oral odor after different interventions.
Oral odor | 1-week after discharge day
  A participant was requested to exhale two gas sampling gas for testing. The investigators uesd an E-nose to identify the participants' odor. To assess the variation of oral odor after different interventions.
Oral odor | 1-month after discharge day
  A participant was requested to exhale two gas sampling gas for testing. The investigators uesd an E-nose to identify the participants' odor. To assess the variation of oral odor after different interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan